CLINICAL TRIAL: NCT06135220
Title: Non-invasive Diagnosis of Pulmonary Embolism by Use of Biomarkers in Exhaled Breath
Acronym: NILEX
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Inger Lise Gade, Principal Investigator, Registrar, MD, PhD, Aalborg University Hospital
Other Study IDs: ILG-PE-2024; 108272 (Other: Den Videnskabsetiske Komite for Region Nordjylland)
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Embolism
Keywords: Breath test; Proteins; Biomarkers
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 1. Exhaled breath
  2. Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- PE confirmed: Patients admitted with confirmed pulmonary embolism.
  Interventions: Diagnostic Test: New method for diagnosis of pulmonary embolism (PE) in order to validate/consolidate 151 putative identified biomarkers for PE in the exhaled breath.
- PE suspected: Patients admitted with suspected, but not confirmed pulmonary embolism.
  Interventions: Diagnostic Test: New method for diagnosis of pulmonary embolism (PE) in order to validate/consolidate 151 putative identified biomarkers for PE in the exhaled breath.
- Controls: Healthy controls - same gender and age (within af range of 10 years) as PE patients.
  Interventions: Diagnostic Test: New method for diagnosis of pulmonary embolism (PE) in order to validate/consolidate 151 putative identified biomarkers for PE in the exhaled breath.

INTERVENTIONS:
Diagnostic Test: New method for diagnosis of pulmonary embolism (PE) in order to validate/consolidate 151 putative identified biomarkers for PE in the exhaled breath. — The collection time will be an average of 7 minutes. As the patient breathes through a mouthpiece, the exhaled breath is lead through the collection device, and an indicative amount af the exhaled air is led into a clear plastic bag. When the plastic bag is fully inflated, it indicates that the minimum required amount of exhaled breath (approximately 30 liters) has passed through the filter.
  Other Names: The exhaled breath will be collected by use of SensAbues which is a commercially available device for the purpose of the collection of proteins from exhaled breath.

SUMMARY:
In this study, a new, non-invasive method for diagnosis of pulmonary embolism (PE) will be tested.

In pre-clinical studies, the investigators have identified 151 putative biomarkers for pulmonary embolism in the exhaled breath, and several of these were also found in a first in-human clinical study what the investigators performed in 2019-2020 (DOI 10.1088/1752-7163/ad0aaa). These biomarkers need consolidation in a clinical setting using an updated collection device and proteomic analysis platform before development of a prototype and further test of this new diagnostic method.

DETAILED DESCRIPTION:
The study will compare the protein profiles of exhaled breath from patients admitted to the Emergency Care Center with suspected pulmonary embolism and controls with same age (within a range of 10 years) and gender. The main-outcome (i.e., means of the relative amounts of specific proteins in the exhaled breath samples) will be compared by unpaired t-tests after assessment of normality and standard deviations within the two groups (PE patients and controls). Furthermore, sensitivity and specificity will be calculated for relevant proteins. The results from analysis of exhaled breath samples from the patients and controls will be compared with results from the porcine model and the first clinical study to confirm and reduce the number of putative biomarkers for PE.

Blood samples (i.e. excess plasma from routine blood samples drawn as a part of routine diagnostic work-up) from the study participants will be stored for standardization of the putative markers and verification and supplementing analysis of the exhaled breath markers. In order to qualify the most suitable markers and substrates for standardization, the analysis of the exhaled breath samples must be completed before the blood samples can be analyzed. Only biochemical, no genetic analysis will be conducted.

ELIGIBILITY:
PE patients:

* Admitted to the Emergency Care Center with suspected PE
* Are conscious and able to understand the given study information.
* Possess legal capacity.
* Age above 18 years.
* Informed, signed consent is obtained.
* Clinically stable, which is defined as patients with stable blood pressure and not in need for other treatments.
* No need for organ support, which comprises need for vasopressors or inotropes, mechanical ventilation, extra corporal circulation, or renal replacement therapy.
* In subjects, where the PE diagnosis is rejected after diagnostic work-up will be included in as clinical controls

Healthy controls:

The healthy age- and gender matched controls will be recruited as a:

• Random sample from the background population who wants to participate voluntarily on a first come, first served basis. They will be recruited from a hospital setting by using posters and by a social media campaign.

Inclusion criteria for healthy controls:

* Same gender and age (within a 10-year range) as an included PE patient.
* Are conscious and able to understand the given study information.
* Possess legal capacity.
* Age above 18 years.
* Informed, signed consent is obtained.

Exclusion criteria for both PE patients and controls:

* Active malignant disease (i.e., ongoing anti-cancer therapy or palliation).
* Current smokers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is expected that 30 patients with confirmed PE, 30 patients with suspected PE, but where diagnostic work-up did not confirm PE and 30 healthy controls will be included in the study over a one-year period.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Amount of exhaled pulmonary embolism-specific proteins | 1-2 years
  The primary outcome is diagnosis of pulmonary embolism by use of one or more novel protein biomarkers in the exhaled breath. The investigators will use semiquantitative analysis to identify the most suitable bomarkers already published: DOI: 10.3390/jcm10215165

CONTACTS AND LOCATIONS:
Overall Officials: Inger L Gade, MD., Ph.D., Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No